CLINICAL TRIAL: NCT04959162
Title: The Effect of Theoretical Knowledge on Resident's Practical Performance in Musculoskeletal Ultrasound- A Randomized Trial
Brief Title: The Effect of Theoretical Knowledge on Resident's Practical Performance in Musculoskeletal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stine Maya Dreier Carstensen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-001
Record Dates: First submitted 2021-07-01; First posted 2021-07-13 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Musculoskeletal Diseases
Keywords: Training; Ultrasound; E-learning
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-learning preparation (Experimental): Will receive e-learning prior to a hands-on course in musculoskeletal ultrasound
  Interventions: Device: E-learning
- Conventional preparation (Active Comparator): Will receive standard information (time, place etc) prior to a hands-on course in musculoskeletal ultrasound
  Interventions: Device: Conventional preparation

INTERVENTIONS:
Device: E-learning — Development of theoretical knowledge using a E-learning platform before attending a hands-on course in musculoskeletal ultrasound
  Arms: E-learning preparation
Device: Conventional preparation — Attending a hands-on course in musculoskeletal ultrasound with no preparation before course start
  Arms: Conventional preparation

SUMMARY:
Musculoskeletal ultrasound( MSUS) is highly operator-dependent and proper training is needed to ensure appropriate use and minimize risk of incorrect image interpretation.To acquire skills in MSUS, it is mandatory to assure training in both the cognitive ability to recognize normal and pathological findings within the images and the psychomotor component of the examination. This study will examine the effect of a novel developed e-learning platform "The Ultrasound LearNing plAtform (ULNA)", on pre- and post-course musculoskeletal ultrasound performance of rheumatology residents. Moreover, to examine the resident's satisfaction with the e-learning platform ULNA.

ELIGIBILITY:
Inclusion Criteria: Residents working in Denmark. Participants are required to have a medical license and provide informed consent before inclusion

Exclusion Criteria:

1. No informed consent
2. Existing The Danish Society for Rheumatology (DRS) level 1 or higher.
3. Participation in prior studies involving musculoskeletal ultrasound training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Difference in The Objective Structures Assessment of Ultrasound skills (OSAUS) score in percent between pre- and post-course assessment for the intervention group and the control group. | 1 year
  Scale (5-25 points). 25 is the maximum score, i.e. the best score

SECONDARY OUTCOMES:
Difference in time used to complete the MSUS examination between the groups. | 1 year

OTHER OUTCOMES:
Comparing the times used on the online platform and the performance score | 1 year
Participant experience using the Intrinsic Motivation Inventory (IMI) scale | 1 year
  Scale (1-7) 1 = not at all true, 7=very true

CONTACTS AND LOCATIONS:
Overall Officials: Stine Maya Carstensen, MD, Principal Investigator — Copenhagen Center for Arthritis Research (COPECARE)
Locations (1):
- COPECARE (Copenhagen Center for Arthritis Research), Glostrup Municipality, Denmark

REFERENCES:
- [Background] Widener BB, Cannella A, Martirossian L, Kissin EY. Modern Landscapes and Strategies for Learning Ultrasound in Rheumatology. Rheum Dis Clin North Am. 2020 Feb;46(1):61-71. doi: 10.1016/j.rdc.2019.09.002. PMID 31757287
- [Background] Carstensen SMD, Terslev L, Jensen MP, Ostergaard M. Future use of musculoskeletal ultrasonography and magnetic resonance imaging in rheumatoid arthritis. Curr Opin Rheumatol. 2020 May;32(3):264-272. doi: 10.1097/BOR.0000000000000709. PMID 32205568
- [Background] Brown AK, Roberts TE, O'connor PJ, Wakefield RJ, Karim Z, Emery P. The development of an evidence-based educational framework to facilitate the training of competent rheumatologist ultrasonographers. Rheumatology (Oxford). 2007 Mar;46(3):391-7. doi: 10.1093/rheumatology/kel415. Epub 2007 Jan 30. PMID 17264091
- [Background] Brown AK, O'Connor PJ, Wakefield RJ, Roberts TE, Karim Z, Emery P. Practice, training, and assessment among experts performing musculoskeletal ultrasonography: toward the development of an international consensus of educational standards for ultrasonography for rheumatologists. Arthritis Rheum. 2004 Dec 15;51(6):1018-22. doi: 10.1002/art.20844. PMID 15593176
- [Background] Kang TL, Berona K, Elkhunovich MA, Medero-Colon R, Seif D, Chilstrom ML, Mailhot T. Web-based teaching in point-of-care ultrasound: an alternative to the classroom? Adv Med Educ Pract. 2015 Mar 13;6:171-5. doi: 10.2147/AMEP.S72159. eCollection 2015. PMID 25792863
- [Background] Filippucci E, Meenagh G, Ciapetti A, Iagnocco A, Taggart A, Grassi W. E-learning in ultrasonography: a web-based approach. Ann Rheum Dis. 2007 Jul;66(7):962-5. doi: 10.1136/ard.2006.064568. Epub 2007 Feb 28. PMID 17329310
- [Derived] Carstensen SMD, Just SA, Velander M, Konge L, Hubel MS, Rajeeth Savarimuthu T, Pfeiffer Jensen M, Ostergaard M, Terslev L. E-learning and practical performance in musculoskeletal ultrasound: a multicentre randomized study. Rheumatology (Oxford). 2023 Nov 2;62(11):3547-3554. doi: 10.1093/rheumatology/kead121. PMID 36943374